CLINICAL TRIAL: NCT06976008
Title: CMV-associated Immunomodulation in Renal Transplant Patients
Acronym: IMMCMV
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: APHP240837; ID-RCB Number : 2024-A01039-38 (Other: France : Ministry of Health)
Record Dates: First submitted 2025-05-09; First posted 2025-05-16 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Kidney Transplantation
Keywords: Kidney transplant; Solid organ transplantation; Cytomegalovirus infection; Immunomodulatory effect of cytomegalovirus infection; Heterologous infection
MeSH Terms: conditions — Cytomegalovirus Infections | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kidney transplant recipients followed since the day of the transplantation (Experimental): Kidney transplant recipients followed since the day of the transplantation
  Interventions: Other: blood sampling
- kidney transplant recipients with CMV viremia (Experimental): kidney transplant recipients with CMV viremia
  Interventions: Other: blood sampling

INTERVENTIONS:
Other: blood sampling — Blood samples will be taken at different timepoints following CMV viremia to evaluate the impact of CMV viremia over time.

SUMMARY:
Cytomegalovirus (CMV) infection has been associated with an increased risk of bacterial, fungal and viral infections in solid organ transplant recipients. The purpose of this study to evaluate if the occurrence of CMV viremia modify the ability to develop optimal immune responses against other pathogens in kidney transplant recipients (heterologous immunity). The objective of this project is to identify the immune pathways affected by CMV in the context of immunosuppression associated with kidney transplantation.

DETAILED DESCRIPTION:
Cytomegalovirus (CMV) infection remains one of the most frequent and problematic complications of solid organ transplantation. Several epidemiological studies have shown an association between CMV infection and the occurrence of severe bacterial or fungal infections. However, the mechanisms by which CMV increases the risk of heterologous infection are still poorly understood. Several data support a direct or indirect immunomodulatory effect of CMV. Indeed, in healthy subjects, CMV seropositivity has a strong phenotypic and functional impact on adaptive immunity while in solid organ transplant patients, a decrease in the innate response to various antigenic stimuli has been observed during CMV viremia. The hypothesis of the study is that the occurrence of CMV viremia reduces the ability to develop optimal immune responses against other targeted pathogens in kidney transplant recipients (heterologous immunity). The objective of this project is to identify the immune pathways affected by CMV in the context of immunosuppression associated with kidney transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. st cohort :

   * Age > 18 years
   * patients with end-stage renal failure programmed for kidney transplantation with a live donor
2. nd cohort :

   * Age > 18 years
   * kidney transplant recipient with CMV viremia

Exclusion Criteria:

- Patients under guardianship, curatorship, legal protection.

For patients with end-stage renal failure scheduled to receive a kidney transplant from a living donor :

* Patients with an active viral (other than CMV), bacterial or fungal infection at the time of inclusion
* patients receiving a desensitization protocol (ABO or anti-HLA)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2029-10-01 (Estimated); Study Completion 2029-10-01 (Estimated)

PRIMARY OUTCOMES:
Impact of CMV infection on the heterologous innate immune response in kidney transplant patients | 12 months
  Comparison of the amount of cytokine production after stimulation of innate immune cells with whole microorganisms (E. Coli, Candida, Aspergillus, influenza virus) in solid organ transplant recipients with and without CMV over time.

SECONDARY OUTCOMES:
Impact of CMV infection on the heterologous adaptive immune response in kidney transplant patients | 12 months
  Comparison of the amount of cytokine production after stimulation of adaptative immune cells with a T-cell superantigen and CMV proteins in solid organ transplant recipients with and without CMV over time.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Serris, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (4):
- France (4):
  - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - Hôpital européen Georges Pompidou, Paris
  - Hôpital Necker-Enfants Malades, Paris
  - Insitut Pasteur, Paris

IPD SHARING:
Plan to Share IPD: No